CLINICAL TRIAL: NCT05195060
Title: The Dutch Cohort Study for the Evaluation of the Use of Neutralizing Monoclonal Antibodies and Other Antiviral Agents Against SARS-CoV-2
Brief Title: TURN-COVID Biobank: The Dutch Cohort Study for the Evaluation of the Use of Neutralizing Monoclonal Antibodies and Other Antiviral Agents Against SARS-CoV-2
Acronym: TURN-COVID
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, W. J. Wiersinga, MD, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL78705.018.21
Record Dates: First submitted 2022-01-07; First posted 2022-01-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — casirivimab; imdevimab; casirivimab and imdevimab drug combination; sotrovimab; molnupiravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma, serum, PBMC's
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19: Patients diagnosed with COVID-19
  Interventions: Drug: casirivimab with imdevimab; Drug: sotrovimab; Drug: molnupiravir

INTERVENTIONS:
Drug: casirivimab with imdevimab — Monoclonal antibody
  Other Names: REGEN-COV
Drug: sotrovimab — Monoclonal antibody
  Other Names: Xevudy
Drug: molnupiravir — antiviral agent
  Other Names: Lagevrio

SUMMARY:
Novel antiviral drugs can mark a turning point in the prevention and treatment of patients with Covid-19. Recently, several independent large phase-III RCTs have shown that the intravenous administration of one gift of neutralizing SARS-CoV-2 monoclonal antibodies can reduce the relative risk of hospital admission and/or death with 70-85% in seronegative patients with SARS-CoV-2 infection when given within 3 to 7 days after state of symptoms. Moreover, novel oral anti-viral compunds such as molnupiravir and nirmatrelvir/ritonavir could reduce the risk of hospitalisation or death by 30% to89% in at-risk adults with Covid-19. These are potential breakthroughs in the treatment of SARS-CoV-2 infection and can be of special importantance for immunocompromised patients who have a diminished or complete lack of an effective humoral response towards Covid-19 vaccination. Monoclonal SARS-CoV-2 antibodies and antivirals have been given an emergency use authorization by regulatory authorities and are or will become available in the Netherlands to treat SARS-CoV-2 infected patients who are at high risk of developing severe disease. Now, urgent key questions need to be addressed: Which patient categories will benefit most from these new drugs? What are the SARS-CoV-2 viral load as well as inflammatory response kinetics during and after treatment with the new SARS-CoV-2 therapies? What is the safety profile in () patients; do new SARS-CoV-2 variants occur during treatment? This study aims to establish a prospective cohort together with a biobank of patients treated with new SARS-CoV-2 therapies to evaluate its real world effect and safety.

Primary Objectives:

* A. What are the SARS-CoV-2 viral load kinetics during and after treatment withneutralizing monoclonal antibodies and other antiviral agents against SARS-CoV-2?
* B. Do viralvariants, spike mutations and immune escape occur during treatment with neutralizing monoclonal antibodies and other antiviral agents against SARS-CoV-2?new SARS-CoV-2 therapies?
* C. What are the viral antibody and inflammatory response kinetics during and after treatment with neutralizing monoclonal antibodies and other antiviral agents against SARS-CoV-2?
* D. To create a biobank to address future questions regarding the current use of neutralizing monoclonal antibodies and other antiviral agents against SARS-CoV-2compared to novel COVID-19 treatments which are in development.

Study design:

Establishment of an observational cohort study including a biobank of patients who receive neutralizing monoclonal antibodies and other novel antiviral agents against SARS-CoV-2.

Study population: All patients above 18 years of age treated with neutralizing monoclonal antibodies and other novel antiviral agents against SARS-CoV-2.

Intervention (if applicable): None Main study parameters/endpoints: Viral load kinetics during treatment. Viral mutations during and after treatment. Presence of monoclonal antibody during treatment and host antibody production and inflammatory responses during treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participating in this observational study will not directly benefit the participants and healthy volunteers. The study will provide information about the effect, host response and safety of thse new anti-SARS-CoV-2 therapies during Covid-19. Clinical data will be obtained through the electronic patient dossier. The knowledge obtained can potentially benefit Covid-19 patients in the future by optimizing treatment strategies. The burden and risks for patients participating in the TURN-COVID biobank study is minimal.

Patients will be visited by a research physician or research nurse during or within three days after receiving neutralizing monoclonal antibodies and other antiviral agents against SARS-CoV-2. Baseline data regarding medical history, admission and vital parameters will be collected through the electronic patient dossier. At the follow-up visits we will draw a total of (3x 43 ML and 1x16 ml = 145 ml of venous blood) and obtain 4 oro-/nasopharyngeal swabs divided over four time-points (day of treatment and day 7, 28 and 90 post treatment).

DETAILED DESCRIPTION:
2. INTRODUCTION AND RATIONALE New SARS-CoV-2 specific monoclonal antibodiestherapies From the beginning of the worldwide pandemic till now no effective specific anti- SARS-CoV-2 treatment was available1,2. In June 2021 the use of SARS-CoV-2 monoclonal antibodies as early treatment for SARS-CoV-2 infected individuals became available in the Netherlands after an emergency use authorisation of the FDA and EMA. First large phase-III randomised controlled clinical trials have showed that SARS-CoV-2 monoclonal antibodies, when given early after the onset of symptoms, bind the SARS-CoV-2 spike protein effectively and prevent hospital admission and death3-7. Additionally, promising SARS-CoV-2 compounds ,such as the oral antivirals molnupiravir8 and nirmatrelvir/ritonavir paxlovid9received recently received an emergency use authorization of the FDA in patients with Covid-19 at high risk of hospitalization and death. EMA's human medicines committee (CHMP) has also started a rolling review of the oral antiviral medicine molnupiravir.

Pathophysiology SARS-CoV-2 monoclonal antibodies

SARS-CoV-2 monoclonal antibodies recognize a single and unique epitope on the SARS-CoV-2 spike proteins and are derived from donor B lymphocytes. The donor B-lymphocytes can be derived either from patients who had Covid-19 or humanized mice who were exposed to SARS-CoV-23,10. The SARS-CoV-2 monoclonal antibodies inhibit the entry of the virus into the host cells (neutralization). Furthermore, antibody binding results in opsonization and is the first step of phagocytosis, eventually resulting in apoptosis and necrosis of the infected cells3. Monoclonal antibodies can be altered artificially in the laboratory to combat emerging variants of SARS-CoV-23. Threewo frequently investigated combinations are casirivimab with imdevimab, sotrovimabsotrovimab and and balanivimab with etesevimab4-7,11.

Small-molecules for Covid-19 At present, many candidate small-molecule therapeutics have been developed that can inhibit both the infection and replication of SARS-CoV-2 and even potentially relieve cytokine storms and other related complications. As SARS-CoV-2 infects cells, reproduces itself, and spreads, the coronavirus relies on dozens of viral and host proteins to complete its life cycle. The new oral pill paxlovid (Phizer) inhibits the main viral protease used to create other proteins for the virus9 (REF. The oral pill molnupiravir (Merck) inserts a defective RNA building block when the virus uses an enzyme known as a polymerase to copy its genome. (REF Molnupiravir)8

The role of SARS-CoV-2new monoclonal antibodies in treatment of SARS-CoV-2 therapies There are a number of factors that most probably will lead to seasonally peaks of infection and hospital admissions for SARS-CoV-2 infections12-14. First, there will remain a group within our population that remains willingly unvaccinated. Second, it is shown that numerous immunocompromised patients have inadequate antibody response to vaccinations and do not produce long-term protection15,16. At last, with new emerging viral variants arising with expected higher viral spread, it is assumed that outbreaks of SARS-CoV-2 infections will remain prevalent in the coming years12-14,17.

With regard to immunocompromised patients, even with the most effective mRNA SARS-CoV-2 vaccines show reduced or even absent humoral responses in patients with solid organ transplants or for instance in patients treated with anti-CD20 for an hematologic malignancy15,16. The fact that immunocompromised patients have inadequate immune response to vaccinations underscores the need of treatment options essential for a subpopulation to slow or stop the replications of the SARS-CoV-2 virus. Especially for these immunocompromised patients the novel neutralizing monoclonal SARS-CoV-2 antibodies therapies could become a real game changer.

First results of phase-III studies SARS-CoV-2 monoclonal antibodies

The first results of three several phase III placebo-controlled randomized controlled clinical trials of monoclonal antibodies of SARS-CoV-2 are now available4,5,7,11. The studies were designed to analyze the effect of these monoclonal antibodies when given early after symptom onset to prevent disease progression, hospital admission and mortality. Although these three studies are currently in pre-print, tTwo other studies recently presented the preplanned interim analysis regarding the treatment of casirivimab with imdevimab4 combination and the sotrovimab alone5. These two studies investigated a single intravenously administration of monoclonal antibodies within 3-7 days after the start of symptoms and demonstrated a relative reduction of 70-85% in Covid-19 related hospital admission and death within four weeks4,18.

Due to the abovementioned evidence, the Dutch medical guideline for the treatment of SARS-CoV-2 patients updated on July 20November, 2021. The Dutch Working Party on Antibiotic Policy (Stichting Werkgroep AntibioticaBeleid, SWAB) now considers to treat patients without a prior antibody response (that means no vaccination response and no seroconversion) and with a high risk of Covid-19 disease progression to start treatment with neutralizing monoclonal SARS-CoV-2 antibodies within 7 days after the start of symptoms19. Patients with a high risk to develop severe Covid-19 are defined as follows in the Dutch guidelines: age > 70 years, medical history of hematologic malignancy in the last five years, severe kidney failure/dialysis, organ or bone marrow transplant, primary immunodeficiency, Downs syndrome, neurologic disease in which the lung ventilation is compromised, body mass index (BMI) >40, or using immunosuppressive medication or age > 60 years in combination with cardiovascular disease, chronic lung/ kidney disease or diabetes 1920.

Before mid December, 2021,At the moment (early Jan 2022), casirivimab plus imdevimab are were the only SARS-CoV-2 monoclonal antibody agents available in the Netherlands. Since then,Of importance however, the B.1.1.529 (Omicron) variant of concern (VOC), which is becoming the dominant variant in many parts ofacross the Netherlands, . This variant, which has numerous mutations in the spike protein, is predicted to have markedly reduced susceptibility to bamlanivimab plus etesevimab and casirivimab plus imdevimab. In line, there is also considerable escape of SARS-CoV-2 Omicron to antibody neutralization by bamlanivimab plus etesevimab. At this moment, sSotrovimab seems to beis the only SARS-CoV-2 monoclonal antibody that is anticipated to have potent neutralisationactivity against the Omicron mutantVOC. Therefore, the Dutch Working Party on Antibiotic adjusted the advice regading the use of casivirmimab plus imdevimab on December 23, 2021. Sotrovimab is expected to become available in the Netherlands in Q1 2022.

Oral SARS-CoV-2 antivirals Small-molecules for Covid-19 The mechanism of action of the nucleoside analogue molnupiravir and the protease inhibitor nirmatrelvir/ritonavir paxlovid areis independent of mutations in the spike protein, which can affect the efficacy of monoclonal antibody treatments. The first results of twoa phase III placebo-controlled randomized controlled clinical trials of molnupiravir oral antivirals for Covid-19 are now available21. are now available. (REF molnupiravir, paxlovid).

Both oral antivirals are developed to be taken within the first few days of Covid-19 infection and are reported expected to reduce the risk of hospitalization and death by approxiametly 30% for molnupiravir and even up tot 89% for nirmatrelvir/ritonavir paxlovid and 30% for molnupiravir.9,21(REF molnupiravir and paxlovid). It should be noted however that compete study results of nirmatrelvir/ritonavir are not yet available. In addition, these compounds were tested in a non-vaccinated population.

The need for an independent Dutch cohort to evaluate the clinical use of neutralizing monoclonalnew SARS-CoV-2 specific antibodiestherapies After the results of these first results of phase-III studies4,5, these compoundsneutralizing monoclonal SARS-CoV-2 antibodies have been given an emergency use authorisation and - since late June 2021 - have become available in the Netherlands to treat SARS-CoV-2 infected patients who are at high risk to develop severe disease. Further randomized controlled trials investigating the effect SARS-CoV-2 antibody in immunocompromised patients are expected to be deemed unethical due to the clear effect seen in the phase-III trials and the already limited existing immune response. Of interest, there are currently only intravenous antibodies treatment regimens available, although the shift to different routes, most notably such as subcutaneous and, intramuscular, oral and inhalation, is underway and will possibly contribute to facilitated and larger access to these monoclonal antibodies. If adequate safety profiles are shown with non-intravenous options a clinical admission could be shortened or prevented. From a safety perspective, it is important to realize that escape by SARS-CoV-2 viral variants have been described from neutralization by convalescent plasma22. Because monoclonal antibodies require administration by means of infusion or injection in a medical setting, oral agents such as molnupiravir and nirmatrelvir/ritonavir paxlovid that can be administered by the patient at home shortly after diagnosis, may be more practical and patient-friendly for nonhospitalized personspatients9,21. As a result, these; such agents are considered would be important new tools in the Covid-19 treatment armamentarium. Another advantage of these oral antivirals over SARS-CoV-2 spike protein-directed monoclonal antibodies is their potential efficacy of against emerging SARS-CoV-2 variants. After the initial results, of the phase III studies (REF paxlovid & molnupiravir), the oral antivirals have been given a FDAn emergency use authorization since late December 2021 by the FDA8,9. Molnupiravir and paxlovid is expected to will become available in the Netherlands in Q1 2022 (nirmatrelvir/ritonavir perhaps in Q2/Q3)February and during the spring, respectively, in the Netherlands. will be available in February and paxlovid in the spring in the Netherlands..

ThisThe above underscores the need to establish a cohort and biobank of patients treated with these compounds in order to monitor this long term outcomes in a real world setting.

Now, urgent key questions need to be addressed to allow the most efficacious use of these novel and potentially lifesaving treatments. Which patient categories will benefit most from these new drugs? What is the safety profile in immunocompromised patients? This study aims to establish a prospective cohort of all patients treated with neutralizing monoclonalnew specific SARS-CoV-2 antibodies therapies to evaluate its real world effect, effect on the host response and safety.

3. OBJECTIVES

Primary Objectives:

To assess effect on the host response and safety of novel SARS-CoV-22 2 monoclonal antibody treatment:therapies.

* A. What are the SARS-CoV-2 viral load kinetics during and after treatment with neutralizing monoclonalnew SARS-CoV-2 antibodiestherapies?
* B. Do SARS-CoV-2 variants, spike mutations and immune escape during treatment with neutralizing monoclonal new SARS-CoV-2 antibodiestherapies?
* C. What are the SARS-CoV-2 antibody and inflammatory response kinetics during and after treatment with neutralizing monoclonalnew SARS-CoV-2 antibodiestherapies?
* D. To create a biobank to address future questions regarding the current use of neutralizing monoclonalnew SARS-CoV-2 antibodies therapies compared to novel COVID-19 treatments which are in development.

  4. STUDY DESIGN

The TURN-COVID biobank will be a prospective cohort study designed in accordance with international standards23. The study population will consist out of all patients treated with monoclonal SARS-CoV-2 antibodies and small-molecules for Covid-19.; this will be primarily patients admitted on the day care facilities for single intravenous dose of neutralizing monoclonal SARS-CoV-2 antibodies but could also include patients that are admitted to the hospital for Covid-19 (see study population). Clinical data will be obtained throughout the electronic patient dossier.

Oropharyngeal swabs and blood samples as detailed below will be sampled at day 0, 7, 28 and 90. A two day deviation before and after the appointment is deemed acceptable for day 0 and day 7. For day 28 and day 90 a seven day deviation is deemed acceptable.. Samples will be stored in the Amsterdam UMC, location AMC. The design is further visualized schematically in Figure 1.

ELIGIBILITY:
Inclusion Criteria:

* All patients that are treated with neutralizing monoclonal SARS-CoV-2 antibodies or with small-molecules for Covid-19 as standard of care.
* Patients have to be aged ≥ 18 y.

Exclusion Criteria:

* No informed consent is provided by the patient or by his/her legal representative
* Patients not suitable to fulfil study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are treated with neutralizing monoclonal SARS-CoV-2 antibodies and with small drug molecules as standard of care for SARS-CoV-2 infection. Patients can receive the intervention in an outpatient setting, ward or ICU. Woman with child bearing potential are included in the study if the treating physician deemed the treatment safe. We will not determine whether or not a a patient receives a treatment as this is the choice of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 1178 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Therapeutic effect of treatment with monoclonal antibodies and antiviral agents | At day 90
Incidence of Treatment-Emergent Adverse Events of treatment with monoclonal antibodies and antiviral agents | At day 90
Cost-effectiveness of treatment with monoclonal antibodies and antiviral agents | At day 90

SECONDARY OUTCOMES:
Change of serologic response during treatment with monoclonal antibodies and antiviral agents | At baseline, day 7, day 28 and day 90

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam University Medical centre - VUMC, Amsterdam, North Holland
  - Amsterdam University Medical Centre, Amsterdam, North Holland
  - Leiden universitair medisch centrum, Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Birnie E, Vergouwe M, Appelman B, Biemond JJ, Heijmans J, Nichols BE, Wiersinga WJ, Popping S; TURN-COVID studygroup. Cost-effectiveness Analysis of Nirmatrelvir/Ritonavir for COVID-19 Among Individuals at High Risk: A Modeling Study. Open Forum Infect Dis. 2025 Mar 26;12(4):ofaf187. doi: 10.1093/ofid/ofaf187. eCollection 2025 Apr. PMID 40256045
- [Result] Vergouwe M, Birnie E, van Veelen S, Biemond JJ, Appelman B, Peters-Sengers H, de Bree GJ, Popping S, Wiersinga WJ; TURN-COVID Study Group. A Longitudinal Description of the Health-Related Quality of Life Among Individuals at High Risk After SARS-CoV-2 Infection: A Dutch Multicenter Observational Cohort Study. Open Forum Infect Dis. 2025 Jan 30;12(2):ofaf055. doi: 10.1093/ofid/ofaf055. eCollection 2025 Feb. PMID 39974282
- [Result] Vergouwe M, Biemond JJ, van der Straten K, van Pul L, Kerster G, Claireaux M, Burger JA, van Dort KA, Kootstra NA, Jonges M, Welkers MRA, Hazenberg MD, Peters-Sengers H, van Gils MJ, Wiersinga WJ, Birnie E, de Bree GJ; TURN-COVID study group. A Robust Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)-Specific T- and B-Cell Response Is Associated With Early Viral Clearance in SARS-CoV-2 Omicron-Infected Immunocompromised Individuals. J Infect Dis. 2024 Oct 16;230(4):e860-e871. doi: 10.1093/infdis/jiae306. PMID 38843052
- [Result] Popping S, Nichols BE, Appelman B, Biemond JJ, Vergouwe M, Rosendaal FR, van der Valk M, de Bree GJ, Wiersinga WJ, Birnie E; TURN-COVID study group. Health Outcomes and Cost-effectiveness of Monoclonal SARS-CoV-2 Antibodies as Pre-exposure Prophylaxis. JAMA Netw Open. 2023 Jul 3;6(7):e2321985. doi: 10.1001/jamanetworkopen.2023.21985. PMID 37410460
- [Result] Birnie E, Biemond JJ, Appelman B, de Bree GJ, Jonges M, Welkers MRA, Wiersinga WJ. Development of Resistance-Associated Mutations After Sotrovimab Administration in High-risk Individuals Infected With the SARS-CoV-2 Omicron Variant. JAMA. 2022 Sep 20;328(11):1104-1107. doi: 10.1001/jama.2022.13854. PMID 35913747